CLINICAL TRIAL: NCT04521166
Title: Investigating the Relationship Between Directional Microphones, Compression, and Working Memory in Realistic Spatial Conditions.
Brief Title: Hearing Aid Processing and Working Memory in Realistic Spatial Conditions
Acronym: DIRWDRCWM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Pamela Souza, Professor, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: STU00210459; K01DC018324 (NIH)
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss, Sensorineural
Keywords: hearing aids; directional microphones; cognition; compression
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Hearing Aids

STUDY DESIGN:
Intervention Model Description: Settings in a wearable hearing aid will be adjusted within a clinically-relevant range for two features. The features include wide dynamic range compression and microphone directionality.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant will be blinded to the hearing aid features being adjusted. The order of presentation of the hearing aid features will be randomized across participants, using a Latin-Square design. The outcomes assessor(s) (who score speech intelligibility) will also be blinded to the conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Setting 1 (Experimental): Hearing aid features presented in this arm include omnidirectional microphone settings and fast-acting compression
  Interventions: Device: Hearing aid
- Setting 2 (Experimental): Hearing aid features presented in this arm include omnidirectional microphone settings and slow-acting compression
  Interventions: Device: Hearing aid
- Setting 3 (Experimental): Hearing aid features presented in this arm include directional microphone settings and fast-acting compression
  Interventions: Device: Hearing aid
- Setting 4 (Experimental): Hearing aid features presented in this arm include directional microphone settings and slow-acting compression
  Interventions: Device: Hearing aid

INTERVENTIONS:
Device: Hearing aid — Settings in a wearable hearing aid will be adjusted within a clinically-relevant range for two features. The features include wide dynamic range compression and microphone directionality.

SUMMARY:
The goal of this project is to determine whether the selection of hearing aid settings should be based in part on an individual's cognitive characteristics (specifically, working memory). We anticipate the outcomes of this study to be applicable to realistic listening conditions.

DETAILED DESCRIPTION:
Hearing aids have specialized features to improve access to sounds for the hearing-impaired listener. The choice of appropriate hearing aid settings is integral to the hearing rehabilitative process. Researchers and clinicians have been influenced by previous work showing that individual cognitive abilities, including working memory, are associated with hearing aid benefit, especially in adverse listening conditions. However, previous research is limited to omnidirectional microphone settings and unrealistic listening conditions. Such conditions fail to recognize that most hearing aids are fit with directional processing that may improve the listening environment, and that typical environments contain speech and noise signals in a range of spatial locations. Therefore, the broad goal of this research is to understand how patient variables interact with hearing aid signal processing in realistic listening conditions in order to effectively treat hearing-impaired individuals in communications situations that are most important to them.

ELIGIBILITY:
Inclusion Criteria:

* > =18 years of age; any sex
* Sensorineural hearing loss with pure-tone thresholds between 25-70 decibel hearing level (dB HL) at octave frequencies between 250 and 3000 Hz
* Speak English as their primary language
* Normal or corrected-to-normal vision (<=20/50)
* Participants will be in good health (self-report)

Exclusion Criteria:

* Clinically significant unstable or progressive medical conditions
* Participants who score < 23 on the cognitive screening test (Montreal Cognitive Assessment)
* Evidence of conductive hearing loss or middle ear issues
* Significant history of otologic or neurologic disorders
* Evidence of significant asymmetry between ears
* Non-English-speaking or non-native English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Varsha Rallapalli, AuD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rallapalli V, Freyman R, Souza P. Relationship Between Working Memory, Compression, and Beamformers in Ideal Conditions. Ear Hear. 2025 Mar-Apr 01;46(2):523-536. doi: 10.1097/AUD.0000000000001605. Epub 2024 Nov 6. PMID 39620655

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the local community in the Chicago area
Groups:
- Hearing Aid Setting: Single Arm: All participants listened to hearing aid features presented in this arm include omnidirectional microphone settings, directional microphone settings, slow-acting compression, and fast-acting compression
  Hearing aid: Settings in a wearable hearing aid will be adjusted within a clinically-relevant range for two features. The features include wide dynamic range compression and microphone directionality.
Period: Sub-study 1
Arm/Group | Hearing Aid Setting: Single Arm
Started | 21
Completed | 21
Not Completed | 0
Period: Sub-study 2
Arm/Group | Hearing Aid Setting: Single Arm
Started | 23 (Participation in Sub-study 2 and Sub-study 3 was optional for the participants from Sub-study 1. Additionally, participants were allowed to participate in any of the Sub-studies independent from other Sub-studies. From Sub-study 1 to Sub-study 2, 7 participants continued, 14 dropped out, 16 were added.)
Completed | 23
Not Completed | 0
Period: Sub-study 3
Arm/Group | Hearing Aid Setting: Single Arm
Started | 17 (Participation in Sub-study 3 was optional for the participants from Sub-study 1 and Sub-study 2. Additionally, participants were allowed to participate in any of the Sub-studies independent from other Sub-studies. From Sub-study 2 to Sub-study 3, 9 participants continued, 14 dropped out, 8 were added. Among the participants added newly in Sub-study 3, there were 3 participants previously completed Sub-study 1 (but not Sub-study 2). Total of 5 participants completed all 3 Sub-studies.)
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants within a Sub-study received all the hearing aid settings. The order of the settings was randomized for each individual participant at the point of testing. Participants were not assigned to a particular order. Participants were allowed to participate in one to three Sub-studies and participation in all Sub-studies was not required.
Groups:
- Hearing Aid Setting: Hearing aid features presented in this arm include omnidirectional microphone settings, directional microphone settings, fast-acting compression, and slow-acting compression
  Hearing aid: Settings in a wearable hearing aid will be adjusted within a clinically-relevant range for two features. The features include wide dynamic range compression and microphone directionality.
Arm/Group | Hearing Aid Setting
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.76 (7.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 42
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 42
Decibel Hearing Level [Mean (Standard Deviation); unit: Decibel Hearing Level] | 38.38 (9.67)
Working Memory Capacity: Percentage of words recalled correctly [Mean (Standard Deviation); unit: Percentage] | 44.16 (11.35)

OUTCOME MEASURES:

1. Primary Outcome: Speech Intelligibility (Percent Correct Scores)
Description: Listeners will listen to and repeat recorded low-context sentences mixed with noise from different spatial locations. Speech intelligibility will be measured immediately following hearing aid fitting. Scoring is determined by percentage of words repeated correctly. Scores range from 0-100% (higher score indicates better performance). This task may take up to 1-2 visits (~ 2 hours each) for different combinations of hearing aid features. The device will only be worn in the laboratory for the duration of the experimental task and will be retrieved by the investigator at the end of each visit.
Time Frame: ~20 mins for each intervention over the course of 1-2 days
Population: A total of 42 participants were tested for the study. The study design was a full factorial design where each participant completed the outcome measures with all 4 settings in sub-studies 1 & 2. In Sub-study 3, the outcome measures were completed with Settings 1 & 3 only. Due to an error in assigning settings, 1 participant each did not listen with settings 1 & 3 in sub-study 1; 1 participant did not listen with Setting 3 in sub-study 3.
Measure: Mean (95% Confidence Interval); unit: percentage of words correct
Units Other Than Participants: Data Points
Arm/Group | Setting 1 | Setting 2 | Setting 3 | Setting 4
Number analyzed (Participants) | 41 | 37 | 40 | 37
Number analyzed (Data Points) | 61 | 43 | 59 | 44
percentage of words correct | 0.55 [0.52 to 0.57] | 0.59 [0.56 to 0.62] | 0.70 [0.67 to 0.73] | 0.80 [0.78 to 0.82]
Statistical Analysis 1: Comparison: Setting 1 vs Setting 2; Test type: Other — A linear mixed model was used to assess whether there was a difference between Settings 1 and 2; p = 0.5291, Mixed Models Analysis — The a priori threshold for statistical significance was 0.05. P-value was adjusted for multiple comparisons using the Bonferroni correction; Slope = -0.00990, 95% CI 2-sided [-0.04075 to 0.02095], Standard Error of Mean 0.01572 — Setting 2 was considered as the reference and the estimate reflects whether the slope for Setting 1 is significantly different from the slope for Setting 2
Statistical Analysis 2: Comparison: Setting 2 vs Setting 3; Test type: Other — A linear mixed model was used to assess whether there was a difference between Setting 2 and Setting 3; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Slope = 0.1329, 95% CI 2-sided [0.09880 to 0.1671], Standard Error of Mean 0.01740 — Setting 2 was considered as the reference and the estimate reflects whether the slope for Setting 3 is significantly different from the slope for Setting 2
Statistical Analysis 3: Comparison: Setting 2 vs Setting 4; Test type: Other — A linear mixed model was used to assess whether there was a difference between Setting 2 and Setting 4; p < .0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Slope = 0.2016, 95% CI 2-sided [0.1660 to 0.2371], Standard Error of Mean 0.01812 — Setting 2 was considered as the reference and the estimate reflects whether the slope for Setting 4 is significantly different from the slope for Setting
Statistical Analysis 4: Comparison: Setting 1; A linear mixed model was used to assess whether there was an effect of working memory on the primary outcome measure (speech intelligibility) after controlling for age and degree of hearing loss (decibel hearing level); Test type: Other — A linear mixed model was used to assess whether there was an effect of working memory on the primary outcome measure (speech intelligibility) after controlling for age and degree of hearing loss (decibel hearing level); p = 0.242, Mixed Models Analysis — The a priori threshold for statistical significance was 0.05; Slope = 0.002
Statistical Analysis 5: Comparison: Setting 2; [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 1, analysis 4]; p = 0.242, Mixed Models Analysis — The a priori threshold for statistical significance was 0.05; Slope = 0.002
Statistical Analysis 6: Comparison: Setting 3; A linear mixed model was used to assess whether there was an effect of working memory on the primary outcome measure (speech intelligibility) after accounting for age and degree of hearing loss (decibel hearing level); Test type: Other — A linear mixed model was used to assess whether there was an effect of working memory on the primary outcome measure (speech intelligibility) after accounting for age and degree of hearing loss (decibel hearing level); p = 0.242, Mixed Models Analysis — The a priori threshold for statistical significance was 0.05; Slope = 0.002
Statistical Analysis 7: Comparison: Setting 4; [analysis description as in outcome 1, analysis 6]; Test type: Other — [test comment as in outcome 1, analysis 6]; p = 0.242, Mixed Models Analysis — The a priori threshold for statistical significance was 0.05; Slope = 0.002

ADVERSE EVENTS:
Time Frame: No adverse events to report because all-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Groups:
- Hearing Aid Setting: Hearing aid features presented in this arm include omnidirectional microphone settings, directional microphone settings, fast-acting compression, and slow-acting compression.
  Hearing aid: Settings in a wearable hearing aid will be adjusted within a clinically-relevant range for two features. The features include wide dynamic range compression and microphone directionality.
Arm/Group | Hearing Aid Setting
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Listeners were tested on the same day as the hearing aid fitting and were not provided with time to acclimate to the different settings. Experience with the different hearing aid settings could affect the role of working memory in speech understanding with hearing aids.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT04521166/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT04521166/SAP_001.pdf